CLINICAL TRIAL: NCT00941213
Title: Comparison of the Quantity of Bleeding and the Duration of Operation in Thoracoscopic Ventral Spondylodesis During Preparation With Monopolar Electrosurgery Compared to Ultrasound Scissors.
Brief Title: Monopolar Electrosurgery Versus Ultrasound Scissors in Thoracoscopic Ventral Spondylodesis
Acronym: Harmonic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Collaborators: Ethicon Endo-Surgery (Europe) GmbH (Industry)
Responsible Party: Dr. med. Peer Eysel, Head of the Department, University of Cologne, Department for Orthopaedics/Trauma Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Uni-Koeln-1235; Uni-Koeln-1235
Record Dates: First submitted 2009-06-15; First posted 2009-07-17 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Fractures of Vertebral Bodies
Keywords: fractures of vertebral bodies Th10-L2; (AO A1 with kyphosis, A2.3, B or C-type)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monopolar Electrosurgery (Active Comparator): Preparation during the operation with Monopolar Electrosurgery
  Interventions: Device: electroscalpel (Erbe Vio 300; Aesculap AG)
- Ultrasound scissors (Experimental): Preparation during the operation with ultrasound scissors
  Interventions: Device: ultrasound scissors - Harmonic ACE

INTERVENTIONS:
Device: ultrasound scissors - Harmonic ACE — preparation with ultrasound scissors during operation
  Other Names: Harmonic ACE; Firma Ethicon Endo-Surgery
  Arms: Ultrasound scissors
Device: electroscalpel (Erbe Vio 300; Aesculap AG) — preparation with electroscalpel during operation
  Other Names: Generator Erbe Vio 300, hook from Aesculap AG
  Arms: Monopolar Electrosurgery

SUMMARY:
This study was undertaken to investigate the effect of using ultrasound scissors in the preparation for Thoracoscopic Ventral Spondylodesis. Quantity of bleeding and the duration of operation in Thoracoscopic Ventral Spondylodesis are compared to the preparation with monopolar electrosurgery.

DETAILED DESCRIPTION:
One group of patients will be operated on using ultrasound scissors in the preparation during Thoracoscopic Ventral Spondylodesis. The other group will be operated on using Monopolar Electrosurgery.

The study is designed as a randomized trial. That means that all patients who have given their consent to participate in the study will be allocated to either ultrasound scissors or Monopolar Electrosurgery by chance.

A total of 40 patients will be included in this study. The study ends with finishing of the first day after the operation, there is no longer follow up.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* fracture of vertebral bodies Th10-L2 with indication for operative treatment

Exclusion Criteria:

* missing informed consent
* mission indication for operative treatment
* revision of the trailing edge
* clotting inhibition therapy
* ASA III/IV
* pregnancy
* malfunction of liver Child C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
duration of the operation | end of the scin suture at the end of operation

SECONDARY OUTCOMES:
loss of blood during operation and at first day after the operation | 24 hours after end of operation
length of stay at the hospital | day of discharge from hospitalization
trauma of internal organs during operation | end of the scin suure at the end of operation

CONTACTS AND LOCATIONS:
Overall Officials: Peer Eysel, Professor, Study Director — University of Cologne, Department of Orthopaedics/Trauma surgery; Gereon Schiffer, MD, Principal Investigator — University of Cologne, Department of Orthopaedics/Trauma surgery
Locations (2):
- Germany (2):
  - University of Cologne, Department of Orthopaedics/Trauma surgery, Cologne, North Rhine-Westphalia
  - Kliniken der Stadt Köln gGmbH Merheim, Cologne, North Rhine-Westphalia